CLINICAL TRIAL: NCT04722939
Title: Identifying Neurocognitive Outcomes and Cerebral Oxygenation in Critically Ill Adults on Acute Kidney Replacement Therapy in the Intensive Care Unit
Brief Title: Neurocognitive Outcomes for ICU Patients With Acute Kidney Injury
Acronym: INCOGNITOAKI
Status: Recruiting | Type: Observational
Sponsor: Dr. Gordon Boyd (Other)
Responsible Party: Sponsor-Investigator, Dr. Gordon Boyd, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-2424-20
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Delirium; Acute Kidney Injury; Critical Illness; Cognitive Impairment; Cerebral Oxygenation; Cerebral Autoregulation
MeSH Terms: conditions — Delirium; Acute Kidney Injury; Critical Illness; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical illness with acute kidney injury: See below for detailed inclusion/exclusion criteria
  Interventions: Diagnostic Test: Cerebral oxygenation

INTERVENTIONS:
Diagnostic Test: Cerebral oxygenation — Cerebral oxygenation will be monitored with the FORESIGHT Elite cerebral oximeter during the first 72h of critical illness, and during subsequent hemodialysis sessions

SUMMARY:
Introduction. Initiation of acute kidney replacement therapy (KRT) is common in critically ill adults admitted to the intensive care unit (ICU), and is associated with increased morbidity and mortality. KRT has been linked to poor neurocognitive outcomes, leading to a reduced quality of life, as well as increased utilization of healthcare resources. Adults initiated on dialysis in the ICU may be particularly at risk of neurocognitive impairment, as survivors of critical illness are already predisposed to developing cerebrovascular disease and cognitive dysfunction over the long-term relative to healthy controls. Regional cerebral oxygen saturation (rSO2) may provide a critical early marker of long-term neurocognitive impairment in patients in this population. The INCOGNITO-AKI study aims to understand cerebral oxygenation in patients undergoing KRT, either continuous or intermittent, in the ICU. These findings will be correlated with long-term cognitive and functional outcomes, as well as structural brain pathology.

Methods and analysis. 108 patients scheduled to undergo treatment for acute kidney injury with KRT in the Kingston Health Sciences Centre ICU will be recruited into this prospective observational study. Enrolled patients will be assessed with intradialytic cerebral oximetry using near infrared spectroscopy (NIRS). Delirium will be assessed daily with the Confusion Assessment Method-Intensive Care Unit (CAM-ICU) and delirium severity quantified as cumulative CAM-ICU-7 scores. Neurocognitive impairment will be assessed at 3- and 12-months after hospital discharge using the Kinarm and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Structural brain pathology on MRI will also be measured at the same timepoints. Driving safety, adverse events, and medication adherence will be assessed at 12-months to evaluate the impact of neurocognitive impairment on functional outcomes.

Ethics and dissemination. This study has been approved by the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board (Approval number: DMED-2424-20). Results will be presented at critical care scientific conferences and a lay summary will be provided to patients and families in their preferred format.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years
* admitted to the Kingston Health Sciences Intensive Care Unit
* diagnosis of severe AKI requiring Kidney Replacement Therapy (KRT) (defined by the presence of either a twofold increase in serum creatinine from baseline, serum creatinine level greater than or equal to 354 micromol/L with an increase of 27 micromol/L from baseline, or urine output <6 mL/kg in the preceding 12 hours)
* within 12 hours of initiation of KRT via intermittent hemodialysis (iHD) or continuous kidney replacement therapy (CKRT).

Exclusion Criteria:

* acquired or congenital neurological disorders
* any contraindication to testing with cerebral oximetry, Kinarm, or MRI (e.g., claustrophobia, limb amputation, paresis, neuromuscular disorders, etc.)
* KRT via PD
* failure to consent
* life expectancy less than 24 hours
* clinical suspicion of renal obstruction
* rapidly progressive glomerulonephritis or interstitial nephritis
* prehospitalization eGFR <30 mL/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Kingston Health Sciences Centre Intensive Care Unit (ICU), which is a 33-bed medical/surgical/trauma/neurological ICU. Patients admitted to the ICU generally require invasive mechanical ventilation for respiratory failure and/or vasoactive medications for hemodynamic support.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Delirium Severity | Patients will be screened daily in the ICU with the CAM-ICU-7 score up until the date of ICU discharge or day 30 of ICU stay.
  Delirium severity will be calculated from the cumulated Confusion Assessment Method-Intensive Care Unit-7 (CAM-ICU-7) score

SECONDARY OUTCOMES:
Cognitive Impairment-Kinarm | 3 months and 12 months
  Patients will undergo a neurocognitive battery with the Kinarm robot and Kinarm standardized tests.
Cognitive Impairment-Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 3 months and 12 months
  Patients will undergo assessment with the RBANS administered by a trained researcher.
Medication adherence | 12 months
  Medication adherence will be assessed with the Medication Adherence Rating Scale (MARS)
Driving safety-1 | 12 months
  Driving safety will be assessed by number of motor vehicle accidents.
Driving safety-2 | 12 months
  Driving safety will be assessed by and the Manchester Driver Behavior Questionnaire
Health care utilization | Within 12 months of hospital discharge.
  We will measure emergency department visits and hospital readmissions.
Structural brain imaging | 3 months and 12 months
  Anonymized and de-identified MRI scans will be processed using MIPAV55 v.7.3.0 and Oxford Centre for Functional MRI of the Brain (FMRIB) Software Library (FSL) v.5.0 medical image processing programs. Scans will be corrected for intensity non-uniformity and transformed into a common image space to adjust for variations in head size and orientation. Skull stripping will be performed. Automated and semi-automated techniques will be used to determine whole-brain volumes from T1-weighted images for analysis of macrostructural brain integrity, as well as FA and MD measures from diffusion-weighted images for analysis of microstructural brain integrity. Brain volumes will be corrected for total intracranial volume to account for head size. Reasons for non-completion of MRI scanning will be recorded. Patients will be used as their own controls over time using a within-subjects design.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individualized patient data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: We are in the final stages of submitting our study protocol for peer review.

REFERENCES:
- [Derived] Jawa NA, Silver SA, Holden RM, Scott SH, Day AG, Norman PA, Kwan BYM, Maslove DM, Muscedere J, Boyd JG. Neurological Impairment in Critically Ill Patients on Dialysis: Research Letter for the INCOGNITO-AKI Feasibility Study. Can J Kidney Health Dis. 2023 Aug 24;10:20543581231192743. doi: 10.1177/20543581231192743. eCollection 2023. PMID 37644980
- [Derived] Jawa NA, Holden RM, Silver SA, Scott SH, Day AG, Norman PA, Kwan BYM, Maslove DM, Muscedere J, Boyd JG. Identifying neurocognitive outcomes and cerebral oxygenation in critically ill adults on acute kidney replacement therapy in the intensive care unit: the INCOGNITO-AKI study protocol. BMJ Open. 2021 Aug 17;11(8):e049250. doi: 10.1136/bmjopen-2021-049250. PMID 34404711